CLINICAL TRIAL: NCT04452110
Title: Investigation of the Reliability of Ultrasonography Usage in the Diagnosis of Temporomandibular Joint Diseases: A Prospective Study
Brief Title: Investigation of the Reliability of Ultrasonography Usage in the Diagnosis of Temporomandibular Joint Diseases
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Ahmet Faruk ERTURK, Principal Investigator, Istanbul University
Other Study IDs: 2019/73; 34908 (Other Grant/Funding Number: Scientific Research Projects Coordination Unit of Istanbul University); 2019-188 (Other: Republic of Turkey Ministry of Health)
Record Dates: First submitted 2020-06-23; First posted 2020-06-30 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Device Reliability
Keywords: Ultrasonography
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I: In volunteers in Group 1, values obtained using a linear probe will be compared.
  Interventions: Diagnostic Test: Ultrasonography
- Group II: In volunteers in Group 2, values obtained using a hockey stick probe will be compared.
  Interventions: Diagnostic Test: Ultrasonography

INTERVENTIONS:
Diagnostic Test: Ultrasonography — Temporomandibular joint diseases of ultrasonography its effectiveness and reliability in diagnosis disadvantages in MR and other imaging methods be ruled out.

SUMMARY:
In the literature, temporomandibular joint diseases on the diagnostic value of the use of ultrasonography in diagnosis studies are lacking. In this study in the diagnosis of temporomandibular joint diseases revealing the reliability of the use of ultrasonography. It is aimed to contribute to the literature in terms of.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 who apply with TMJ problems
* Patients with pain in the joint and chewing muscle area

Exclusion Criteria:

* Syndromic patients
* Patients under the age of 18
* Patients with a history of orthognathic surgery
* Pregnants
* Antidepressant Users
* Patients Using Removable Dentures
* Patients who have had joint treatment in the past six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients Applying to Our University
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Joint Pain Scale | 1 year
  Research Diagnostic Criteria for Temporomandibular Disorders (RDC/TMD) form will be used in our study

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Dentistry Faculty, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Erturk AF, Yelken Kendirci M, Ozcan I, Gokcen Rohlig B. Use of ultrasonography in the diagnosis of temporomandibular disorders: a prospective clinical study. Oral Radiol. 2023 Apr;39(2):282-291. doi: 10.1007/s11282-022-00635-w. Epub 2022 Aug 3. PMID 35920968

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-09): https://cdn.clinicaltrials.gov/large-docs/10/NCT04452110/Prot_SAP_000.pdf
  • Informed Consent Form (2019-09-09): https://cdn.clinicaltrials.gov/large-docs/10/NCT04452110/ICF_001.pdf